CLINICAL TRIAL: NCT00503399
Title: Comparison of the Effects of Teriparatide With Those of Risedronate on Lumbar Spine vBMD in Glucocorticoid-Induced Osteoporosis in Men
Brief Title: Comparison of the Effects of 2 Drugs on Lumbar Spine Volumetric BMD in Men With Glucocorticoid-Induced Osteoporosis
Acronym: EuroGIOPS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11716; B3D-EW-GHDH (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-07-16; First posted 2007-07-18 (Estimated); Results first posted 2011-11-08 (Estimated); Last update posted 2012-03-13 (Estimated); Status verified 2011-10

CONDITIONS: Osteoporosis
Keywords: Glucocorticoid Induced
MeSH Terms: conditions — Osteoporosis | interventions — Teriparatide; Risedronic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Teriparatide (Experimental): Teriparatide 20 microgram (µg) subcutaneous (sc) injection once daily (QD).
  Interventions: Drug: Teriparatide
- Risedronate (Active Comparator): Risedronate 35 milligrams (mg) oral (po) tablet once weekly (QW)
  Interventions: Drug: Risedronate

INTERVENTIONS:
Drug: Teriparatide — 20 µg/day sc for 18 months
  Other Names: LY333334; Forteo; Forsteo
  Arms: Teriparatide
Drug: Risedronate — 35 mg/week po for 18 months
  Other Names: Actonel
  Arms: Risedronate

SUMMARY:
The objective of this study is to test the hypothesis that teriparatide is superior to the active comparator in the change from baseline to 18 months of lumbar spine volumetric trabecular bone mineral density (BMD) in males with glucocorticoid-induced osteoporosis.

DETAILED DESCRIPTION:
This study is a multinational, European, multicenter, randomized, open-label, active comparator controlled study with 2 study periods: a screening phase of up to 6 weeks, and an open-label treatment phase of 18 months. Approximately 100 adult men with osteoporosis associated with sustained glucocorticoid therapy will be enrolled into the study. Approximately one-half of the participants (at all investigational sites) will be randomized to teriparatide 20 micrograms/day (ug/day given as a subcutaneous (sc) injection), and the other half randomized to risedronate 35 milligrams (mg) once weekly (QW) oral (po) tablet. All participants will receive approximately 1000 mg/day elemental calcium and 800 to 1200 international units per day (IU/day) of vitamin D.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory men 25 years of age and older presenting to Visit 1 with a bone mineral density (BMD) of at least 1.5 standard deviation (SD) below the corresponding normal young adult men average BMD (T score of -1.5 or lower), as determined from the manufacturer's database at any of the following regions of interest: total hip, femoral neck, or lumbar spine
* Have received glucocorticoid therapy at an average dose of at least 5.0 milligrams (mg) per day of prednisone or its equivalent for a minimum of 3 consecutive months immediately preceding screening (Visit 1), as determined by medical history.
* A minimum of 2 lumbar vertebrae (L) in the L-1 through L-3 region must be evaluable by quantitative computerized tomography.
* Normal or clinically insignificant abnormal laboratory values (as determined by the investigator) including serum calcium, parathyroid hormone (PTH) (1 84), and 25 hydroxyvitamin D concentrations, and alkaline phosphatase activity.

Exclusion Criteria:

* Presence of a mild, moderate, or severe spinal fracture in both the twelfth thoracic vertebra (T-12) and first lumbar vertebra (L-1), as determined by the central reading facility using the semiquantitative technique.
* Abnormal albumin-corrected serum calcium levels
* History of unresolved skeletal diseases that affect bone metabolism other than glucocorticoid-induced osteoporosis
* History of malignant neoplasms in the 5 years prior to Visit 2, with the exception of superficial basal cell or squamous cell carcinomas of the skin that have been definitively treated. Increased baseline risk of osteosarcoma; this includes patients with Paget's disease of the bone, previous primary skeletal malignancy, or skeletal exposure to therapeutic irradiation.
* Abnormal thyroid function not corrected by therapy
* Past and/or current treatment with certain medications.

Min Age: 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2007-07; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (13):
- Germany (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bad Nauheim
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frankfurt
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heinsberg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leverkusen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Magdeburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Potsdam
- Greece (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kifissia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thessaloniki
- Italy (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Siena
- Spain (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid

REFERENCES:
- [Derived] Gluer CC, Marin F, Ringe JD, Hawkins F, Moricke R, Papaioannu N, Farahmand P, Minisola S, Martinez G, Nolla JM, Niedhart C, Guanabens N, Nuti R, Martin-Mola E, Thomasius F, Kapetanos G, Pena J, Graeff C, Petto H, Sanz B, Reisinger A, Zysset PK. Comparative effects of teriparatide and risedronate in glucocorticoid-induced osteoporosis in men: 18-month results of the EuroGIOPs trial. J Bone Miner Res. 2013 Jun;28(6):1355-68. doi: 10.1002/jbmr.1870. PMID 23322362
- [Derived] Graeff C, Marin F, Petto H, Kayser O, Reisinger A, Pena J, Zysset P, Gluer CC. High resolution quantitative computed tomography-based assessment of trabecular microstructure and strength estimates by finite-element analysis of the spine, but not DXA, reflects vertebral fracture status in men with glucocorticoid-induced osteoporosis. Bone. 2013 Feb;52(2):568-77. doi: 10.1016/j.bone.2012.10.036. Epub 2012 Nov 10. PMID 23149277
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 174 participants who were enrolled into the study, 92 were eligible and randomly assigned to the treatment arms.
Period: Overall Study
Arm/Group | Teriparatide | Risedronate
Started | 45 | 47
Completed | 38 | 39
Not Completed | 7 | 8
Not completed — Death | 2 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Adverse Event | 0 | 3
Not completed — Lost to Follow-up | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Teriparatide | Risedronate | Total
Number analyzed (Participants) | 45 | 47 | 92
Age Continuous [Mean (Standard Deviation); unit: years] | 57.5 (12.80) | 55.1 (15.54) | 56.3 (14.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 45 | 47 | 92
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 44 | 46 | 90
  Hispanic | 0 | 1 | 1
  East Asian | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  Germany | 19 | 21 | 40
  Greece | 6 | 6 | 12
  Italy | 5 | 8 | 13
  Spain | 15 | 12 | 27
Number of participants with fractures before study [Number; unit: participants]
  With fractures | 19 | 17 | 36
  Without fractures | 26 | 30 | 56

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Lumbar Spine Volumetric Trabecular Bone Mineral Density (BMD) by Quantitative Computerized Tomography (QCT) at 18 Months
Description: Least Squares (LS) Means were adjusted for age, baseline serum aminoterminal propeptide of Type I procollagen (P1NP), fracture less than 12 months before study start, duration of prior bisphosphonate use, screening glucocorticoid dose, and cumulative glucocorticoid dose before and during the trial.
Time Frame: Baseline, 18 months
Population: The analysis population was the primary efficacy population, which included all randomized participants who received at least 1 dose of study medication (full analysis set) and had a lumbar spine volumetric trabecular BMD measurement at baseline and at ≥1 post-baseline visit.
Measure: Least Squares Mean (Standard Error); unit: milligram per cubic centimeter (mg/cm^3)
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 39 | 40
milligram per cubic centimeter (mg/cm^3) | 12.28 (3.16) | 2.94 (3.14)

2. Secondary Outcome: Change From Baseline in Lumbar Spine Volumetric Trabecular Bone Mineral Density (BMD) by Quantitative Computerized Technology (QCT) at 6 Months
Description: Least Squares (LS) Means were adjusted for age, baseline propeptide of Type I procollagen (P1NP), fracture less than 12 months before study start, duration of prior bisphosphonate use, screening glucocorticoid dose, and cumulative glucocorticoid dose before and during the trial.
Time Frame: Baseline, 6 months
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: milligram per cubic centimeter (mg/cm^3)
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 39 | 40
milligram per cubic centimeter (mg/cm^3) | 4.31 (3.15) | 2.52 (3.16)

3. Secondary Outcome: Change From Baseline in High Resolution Quantitative Computerized Technology (HR-QCT) of Integral and Trabecular Bone Mineral Density (BMD) of the 12th Thoracic Vertebra (T12) at 6 Months and 18 Months
Description: Three-dimensional (3-D) microstructure variables of T12 were assessed by HR-QCT. In contrast with regular QCT that assessed 3 millimeter (mm) slide thickness, HR-QCT used segmentation of 1 single vertebra with approximately 100 consecutive slides reconstructed at 300-400 micrometer (µm) slice increments covering the complete vertebral body. Least Squares (LS) Means were adjusted for age, baseline P1NP, fracture less than 12 months before study start, duration of prior bisphosphonate use, screening glucocorticoid dose, and cumulative glucocorticoid dose before and during the trial.
Time Frame: Baseline, 6 months, 18 months
Population: The analysis population was the full analysis set (FAS), which included all randomized participants who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: milligram per cubic centimeter (mg/cm^3)
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 39 | 40
milligram per cubic centimeter (mg/cm^3)
  Integral BMD at 6 months | -0.42 (6.42) | -1.91 (7.11)
  Integral BMD at 18 months | 10.72 (6.22) | 0.68 (7.08)
  Trabecular BMD at 6 months | -0.70 (5.26) | -0.87 (5.85)
  Trabecular BMD at 18 months | 9.53 (5.09) | 0.22 (5.82)

4. Secondary Outcome: Change From Baseline in Anterior Bending and Axial Torsion by Finite Element Analysis in the 12th Thoracic Vertebra (T12) at 6 Months and 18 Months: Stiffness and Strength
Description: Anterior bending and axial torsion were measured using HR-QCT-based finite element analysis to determine stiffness and strength of T12. Stiffness evaluated strength of the vertebral body, defined as the slope of the initial step of the force-displacement curve. Strength of the vertebral body was evaluated under compressive loading conditions using computer simulation. LS Means were adjusted for age, baseline P1NP, fracture less than 12 months before study start, duration of prior bisphosphonate use, screening glucocorticoid dose, and cumulative glucocorticoid dose before and during the trial.
Time Frame: Baseline, 6 months, 18 months
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Newton/millimeter/radian (N/mm/rad)
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 39 | 40
Newton/millimeter/radian (N/mm/rad)
  Anterior bending stiffness at 6 months | 664969.0 (317684.0) | 415705.0 (323135.0)
  Anterior bending stiffness at 18 months | 1209225.0 (300977.0) | 233283.0 (322829.0)
  Axial torsion stiffness at 6 months | 142902.9 (71714.2) | 77830.7 (72947.9)
  Axial torsion stiffness at 18 months | 279392.8 (68284.5) | 56639.3 (72946.9)
  Anterior bending strength at 6 months | 12490.9 (8405.0) | 8827.2 (8741.0)
  Anterior bending strength at 18 months | 26046.4 (8304.1) | 4822.0 (8686.6)
  Axial torsion strength at 6 months | 6127.7 (4132.3) | 3664.0 (4233.5)
  Axial torsion strength at 18 months | 14181.3 (3954.4) | 2545.8 (4228.7)

5. Secondary Outcome: Change From Baseline in Axial Compression by Finite Element Analysis in the 12th Thoracic Vertebra (T12) at 6 Months and 18 Months: Stiffness and Strength
Description: Axial compression was measured using HR-QCT-based finite element analysis to determine stiffness and strength of T12. Stiffness evaluated the strength of the vertebral body, defined as the slope of the initial step of the force-displacement curve. Strength of the vertebral body was evaluated under compressive loading conditions using computer simulation. LS Means were adjusted for age, baseline P1NP, fracture less than 12 months before study start, duration of prior bisphosphonate use, screening glucocorticoid dose, and cumulative glucocorticoid dose before and during the trial.
Time Frame: Baseline, 6 months, 18 months
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Newton per millimeter (N/mm)
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 39 | 40
Newton per millimeter (N/mm)
  Axial compression stiffness at 6 months | 890.7 (596.6) | 407.6 (607.6)
  Axial compression stiffness at 18 months | 1973.9 (569.0) | 363.7 (605.9)
  Axial compression strength at 6 months | 580.7 (444.6) | 313.6 (457.0)
  Axial compression strength at 18 months | 1287.5 (424.0) | 209.4 (455.5)

6. Secondary Outcome: Change From Baseline in Areal Bone Mineral Density (BMD) at Lumbar Spine, Femoral Neck, and Total Hip at 18 Months
Description: Dual x-ray absorptiometry (DXA) techniques validated this measurement at skeletal sites that are at risk of osteoporotic fracture, such as lumbar spine, femoral neck, and hip.
Time Frame: Baseline, 18 months
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: grams per square centimeter (g/cm^2)
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 45 | 47
grams per square centimeter (g/cm^2)
  Lumbar spine (n=38; n=39) | 0.068 (0.0685) | 0.037 (0.0493)
  Hip (n=38; n=37) | 0.014 (0.0319) | 0.007 (0.0320)
  Femoral neck (n=38; n=37) | 0.014 (0.0446) | -0.007 (0.0333)

7. Secondary Outcome: Change From Baseline in Serum Aminoterminal Propeptide of Type I Procollagen (P1NP) at 3 Months, 6 Months, and 18 Months
Description: P1NP was used as a serum biochemical marker of collagen synthesis, reflecting the formation of new osteoid.
Time Frame: Baseline, 3 months, 6 months, 18 months
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: micrograms per deciliter (μg/dL)
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 45 | 47
micrograms per deciliter (μg/dL)
  P1NP at 3 months | 27.33 (8.32) | -16.09 (7.82)
  P1NP at 6 months | 52.55 (8.27) | -16.50 (7.95)
  P1NP at 18 months | 28.48 (8.74) | -15.58 (8.58)

8. Secondary Outcome: Change From Baseline in Serum Type I Collagen Degradation Fragments (β-CTx) at 3 Months, 6 Months, and 18 Months
Description: β-CTx was used as a biochemical marker of bone turnover/resorption, reflecting collagen breakdown of the bone matrix.
Time Frame: 3, 6, 18 months
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: nanograms per deciliter (ng/dL)
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 45 | 47
nanograms per deciliter (ng/dL)
  β-CTx at 3 months | 0.12 (0.07) | -0.15 (0.07)
  β-CTx at 6 months | 0.25 (0.07) | -0.14 (0.07)
  β-CTx at 18 months | 0.03 (0.08) | -0.11 (0.07)

9. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: Summary tables of serious AEs (SAEs) and all other non-serious AEs are located in the Reported Adverse Event Module. Fractures that occurred during the study were collected separately as an additional safety variable. The number of participants experiencing hypercalcemia was summarized for each treatment arm. Hypercalcemia was defined as a serum calcium level corrected for albumin of >2.7 millimole per liter (mmol/L) (10.8 milligram per deciliter [mg/dL]).
Time Frame: Baseline up to 18 months
Population: The safety analysis set included all participants who received study treatment.
Measure: Number; unit: participants
Arm/Group | Teriparatide | Risedronate
Number analyzed (Participants) | 45 | 47
participants
  Serious Adverse Events (SAEs) | 13 | 22
  Other Non-serious AEs | 22 | 30
  Fractures | 0 | 5
  Hypercalcemia | 0 | 0

ADVERSE EVENTS:
Arm/Group | Teriparatide | Risedronate
Serious Adverse Events (participants affected / at risk) | 13/45 | 22/47
Other Adverse Events (participants affected / at risk) | 22/45 | 30/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teriparatide (N=45) | Risedronate (N=47)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1)
Sudden hearing loss (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 1 (2)
Crohn's disease (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Sudden death (General disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Anal abscess (Infections and infestations) | 0 (0) | 1 (1)
Cytomegalovirus infection (Infections and infestations) | 1 (1) | 0 (0)
Intervertebral discitis (Infections and infestations) | 0 (0) | 1 (1)
Postoperative abscess (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (4)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Seminoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Leukoplakia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Scar (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Femoral artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 0 (0) | 2 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Teriparatide (N=45) | Risedronate (N=47)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Reflux oesophagitis (Gastrointestinal disorders) | 1 (1) | 2 (2)
Oedema peripheral (General disorders) | 3 (4) | 2 (2)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Influenza (Infections and infestations) | 4 (4) | 3 (4)
Lung infection (Infections and infestations) | 0 (0) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (2) | 2 (2)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (4)
Blood cholesterol increased (Investigations) | 0 (0) | 2 (2)
Weight decreased (Investigations) | 0 (0) | 2 (2)
Weight increased (Investigations) | 1 (1) | 3 (3)
Obesity (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Headache (Nervous system disorders) | 1 (1) | 2 (3)
Paraesthesia (Nervous system disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Erythema (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Cataract operation (Surgical and medical procedures) | 2 (2) | 1 (2)
Haematoma (Vascular disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days